CLINICAL TRIAL: NCT05183880
Title: Investigating the Oral Bioavailability of Vitamin C Administered Using Phosphycell™ Technology - a Phosphatidylcholine-lipid Encapsulation Technology.
Brief Title: Bioavailability of Orally Ingested Vitamin C
Acronym: ABBA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Vitamin C formulation no longer in production
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 21-10-20-B-01
Record Dates: First submitted 2021-12-21; First posted 2022-01-11 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crystalline vitamin C supplementation (Active Comparator): 1000 mg of vitamin C ingested in crystalline form
  Interventions: Dietary Supplement: Crystalline vitamin C
- Phosphatidylcholine-lipid encapsulated vitamin C supplementation (Experimental): 1000 mg of vitamin C ingested in phosphatidylcholine-lipid encapsulated form
  Interventions: Dietary Supplement: Phosphatidylcholine-lipid encapsulated vitamin C

INTERVENTIONS:
Dietary Supplement: Phosphatidylcholine-lipid encapsulated vitamin C — Ingesting 1000 mg of vitamin C in phosphatidylcholine-lipid encapsulated form
  Arms: Phosphatidylcholine-lipid encapsulated vitamin C supplementation
Dietary Supplement: Crystalline vitamin C — Ingesting 1000 mg of vitamin C in crystalline form
  Arms: Crystalline vitamin C supplementation

SUMMARY:
The purpose of this study is to determine if crystalline vitamin C supplementation can acutely increase skeletal muscle vitamin C concentrations and if this can be potentiated by administering vitamin C using Phosphycell™ Technology - a phosphatidylcholine-lipid encapsulation technology.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) 18.5 - 30 kg/m2
* Age 18 - 40
* Non-smoker

Exclusion Criteria:

* Body mass index (BMI) < 18.5 or > 30 kg/m2
* Age < 18 or > 40
* Smoking
* Cardiovascular disease
* Hypertension (≥ 140/90 mmHg)
* Metabolic disease
* Medications known to affect vitamin C metabolism
* A known vitamin C deficiency
* Less than 2 hours per week of physical activity or following a structured exercise training program.
* Routine use of vitamin supplements

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11-26 (Actual); Primary Completion 2022-11-26 (Estimated); Study Completion 2023-11-26 (Estimated)

PRIMARY OUTCOMES:
Skeletal muscle vitamin C concentrations | 6 hours after vitamin C ingestion
  Skeletal muscle vitamin C concentrations 6 hours after vitamin C ingestion will be measured using HPLC and compared to baseline
Skeletal muscle vitamin C concentrations | 12 hours after vitamin C ingestion
  Skeletal muscle vitamin C concentrations 12 hours after vitamin C ingestion will be measured using HPLC and compared to baseline and 6 hours after vitamin C ingestion

SECONDARY OUTCOMES:
Blood plasma vitamin C concentrations | 24 hours after vitamin C ingestion
  Blood plasma vitamin C concentrations will be measured using HPLC during the 24 hour post vitamin C ingestion period
White blood cell vitamin C concentrations | 6 hours after vitamin C ingestion
  White blood cell vitamin C concentrations will be measured 6 hours after vitamin C ingestion using HPLC and compared to baseline
White blood cell vitamin C concentrations | 24 hours after vitamin C ingestion
  White blood cell vitamin C concentrations will be measured 24 hours after vitamin C ingestion using HPLC and compared to baseline and 3 hours post vitamin C ingestion
Cardiovascular function | 24 hours after vitamin C ingestion
  Cardiovascular function will be measuring using a finger plethysmograph during the 24 hour post vitamin C ingestion period

CONTACTS AND LOCATIONS:
Overall Officials: Francis Stephens, Principal Investigator — University of Exeter
Locations (1):
- Sport and Health Sciences, Exeter, Devon, United Kingdom